CLINICAL TRIAL: NCT00995046
Title: Optimizing Prophylaxis in Patients With Severe Haemophilia A by Tailoring the Infusions to Individual Patients' Needs Using the Calibrated Automated Thrombin Generation Test
Brief Title: Individually Tailored Prophylaxis in Patients With Severe Hemophilia A
Acronym: OPTIPHASE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 2007.482
Record Dates: First submitted 2009-10-12; First posted 2009-10-14 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2009-10

CONDITIONS: Hemophilia A
Keywords: Hemophilia A; prophylaxis; thrombin generation test (TGT)
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- usual prophylaxis regimen (Active Comparator): All patients will receive their usual prophylaxis regimen during the first 6 months
  Interventions: Drug: FVIII
- individually tailored prophylaxis regimen (Experimental): All patients will receive an individually tailored prophylaxis regimen in accordance with TGT results during the second 6 month-period.
  Interventions: Drug: FVIII

INTERVENTIONS:
Drug: FVIII — 6 months of prophylaxis treatment administered 3 or 4 times weekly according to patient's initial regimen, (standardized Malmö protocol 25 - 40 IU/kg/infusion). Medical visits will occur at 3-month intervals (+ 5 days) until the end of the study. Weekly, telephone calls to the patients (parents) will also be done.
  Arms: usual prophylaxis regimen
Drug: FVIII — 1 month period where thrombin generating capacity will be evaluated, followed by 6 months of "individually" tailored prophylaxis regimen according to TGT results. Medical visits will occur at 3-month intervals (+ 5 days) until the end of the study. Weekly, telephone calls to the patients (parents) will also be done.
  Arms: individually tailored prophylaxis regimen

SUMMARY:
Patients with severe haemophilia A lack clotting factor FVIII and suffer from spontaneous and traumatic bleeds. In the absence of treatment, frequent bleeds in joints lead to severe joint destruction. In 1960s, prophylactic therapy was developed involving the infusion of clotting factor on a regular schedule in order to keep clotting levels sufficiently high to prevent spontaneous bleeding episodes. Prophylaxis is started at an early age before the age of 2 years or after the first joint bleed. The Malmö experience indicates that treatment is most effective when administered in large doses at least 3 times weekly. However, such an intensive treatment in young boys may be very difficult to carry out for home treatment. Currently, there is no international recommendation on prophylactic therapy regimens. Because of the high cost and limited availability of factor concentrates, dosing is an important issue in prophylaxis therapy. It was recently shown that 24 hours after FVIII concentrate administration, in patients presenting similar FVIIII levels, thrombin generation capacity may be significantly different. In addition, independently of the FVIII level, a correlation was found between severe clinical bleeding phenotype and thrombin generating capacity. The aim of the present clinical study is to assess the thrombin generation test as the main surrogate marker to evaluate the coagulating capacity of haemophiliacs on prophylaxis regimen. Optimizing prophylactic therapy to patient's phenotype with no loss of clinical effectiveness can significantly improve patients' quality of life, protect haemophilic children against arthropathy and possibly limit the cost of the prophylaxis therapy.

ELIGIBILITY:
Inclusion Criteria:

* Severe haemophilia A (FVIII < 1 IU/dl)
* Currently on prophylactic therapy administered at least 3 times per week with a clinical efficiency
* Age: 6 - 45 years
* Adequate venous access in adults and children i.e. presence of 2 or more good quality peripheral veins, in order to avoid the need for a central venous device. One peripheral vein for FVIII infusions and one other for blood sampling are required.
* Competent in home treatment and infusion therapy (patient or parents)
* Ability of patient or family (for minors) to give informed consent
* Patient affiliated to French Social Insurance System.

Exclusion Criteria:

* Age < 6 years and > 45 years
* Hemophilia A with documented history of inhibitor
* Clinically symptomatic liver disease (supported by e.g. diagnosis of cirrhosis, portal hypertension, ascites, PT > 5 seconds above upper limit of normal)
* Platelet count < 100x109/l
* Planned elective surgery within 13 months
* Poor venous access according inclusion criteria
* Presence of a documented target joint

Ages: 6 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2009-09; Primary Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Consumption of clotting factor concentrate | 13 months

SECONDARY OUTCOMES:
Number of spontaneous bleeds | 13 months
Number of spontaneous joint bleeds | 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Yesim Dargaud, MD, PhD, Principal Investigator — Hospices Civils de Lyon, France
Locations (1):
- Hopital Edouard Herriot, Lyon, France